CLINICAL TRIAL: NCT04126018
Title: Assessment of Left Ventricular Volumes and Strain and Assessment of Valvular Lesions Using Two- and Three-dimensional Echocardiography and Cardiac MRI, a Correlation Study
Brief Title: Comparative Imaging Assessment of Valvular Heart Disease
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Deborah Kwon, MD, Principal Investigator, The Cleveland Clinic
Other Study IDs: 19-549
Record Dates: First submitted 2019-08-20; First posted 2019-10-14 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Valve Heart Disease; Aortic Stenosis; Aortic Regurgitation
MeSH Terms: conditions — Heart Valve Diseases; Aortic Valve Stenosis; Aortic Valve Insufficiency | interventions — Magnetic Resonance Imaging; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — As part of an optional sub study, subjects will be asked to provide blood samples at the baseline visit. Up to 5 tablespoons (75ml) of blood will be drawn. Genomic analyses will be run on the samples to look for biomarkers which may correlate with the development of myocardial fibrosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Mitral Valve Regurgitation: Patients with moderate or severe (3+ or 4+) mitral valve regurgitation on the basis of prior known clinical history or clinical exam.
  Interventions: Diagnostic Test: MRI with strain measurement; Diagnostic Test: Echocardiography
- Aortic Valve Regurgitation: Patients with moderate or severe (3+ or 4+) aortic valve regurgitation on the basis of prior known clinical history or clinical exam.
  Interventions: Diagnostic Test: MRI with strain measurement; Diagnostic Test: Echocardiography
- Aortic Stenosis: Patients with moderate or severe (3+ or 4+) aortic stenosis on the basis of prior known clinical history or clinical exam.
  Interventions: Diagnostic Test: MRI with strain measurement; Diagnostic Test: Echocardiography
- Patients referred for CRT Implantation: Patients who meet clinical guideline criteria for CRT implantation with EF < 40%
  Interventions: Diagnostic Test: MRI with strain measurement; Diagnostic Test: Echocardiography

INTERVENTIONS:
Diagnostic Test: MRI with strain measurement — CMR measurements of left and right ventricular systolic function strain and myocardial fibrosis
Diagnostic Test: Echocardiography — Doppler, PISA, VCA, volumetric method as performed during echocardiography

SUMMARY:
The purpose of the study is to compare the various 2D and 3D methods of valvular heart disease quantification (Doppler, PISA, VCA, volumetric method) and strain with cardiac magnetic resonance (CMR) measurements of left and right ventricular systolic function strain and myocardial fibrosis assessment.

DETAILED DESCRIPTION:
The objective of this study is to compare the accuracy of 3D TTE to 2D TTE in assessing the severity of valvular heart disease in patients with aortic stenosis, aortic regurgitation, and mitral valve regurgitation by comparing this to the reference standard of cardiac magnetic resonance (CMR) in subjects with different etiologies and mechanisms of valvular lesions and to the integrative method of valvular lesion grading as recommended by inter-societal guidelines. Another objective is to assess prevalence of focal and diffuse myocardial fibrosis as assessed by CMR in patients with aortic stenosis, aortic regurgitation and mitral regurgitation. In addition, the investigators aim to determine whether severity of myocardial fibrosis predicts onset of symptoms, referral for valve surgery and adverse ventricular remodeling. The investigators also aim to look at patients who will be undergoing CRT implant to predict their response to therapy.

At baseline, the Rapid Assessment of Physical Activity questionnaire and the Kansas City Cardiomyopathy Questionnaire will be completed. A 6-12 month follow-up is required and will include an abbreviated non-contrast research cardiac MRI and subject questionnaires.

Other follow-up will include using electronic medical records and the Social Security Death Index database for outcomes such as death, hospitalization for heart failure, mitral or aortic valve interventions and cardiovascular death.

Select patients will be asked to undergo a supine bicycle exercise stress MRI at enrollment. Approximately 40 subjects will be included in this substudy.

Additional exclusion criteria for this substudy:

* Unable to pedal a supine bicycle
* Require supplemental oxygen

During the exercise stress MRI, patients will be asked to cycle on a supine bike that will be mounted on the MRI platform. During this test, a caregiver will be present. An electrocardiogram (ECG) will be used to obtain tracings of cardiac activity. Respirations, blood pressure, and heart rate are also monitored during exercise. The test is continued until peak exercise level or target heart rate is achieved. As soon as the exercise portion is complete, MRI images will be acquired. When the test is complete, patients will be monitored until ECG, heart rate, and breathing have returned to baseline. Patients will be assessed for symptoms such as chest pain, dyspnea, leg pain, dizziness, or fatigue and may be given medications or instructed to stop the test early as necessary.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90 years of age
* Suspected moderate or severe MR,AR or AS on the basis of prior known clinical history or clinical exam.
* Suspected CRT "non-responder" with an implanted MRI compatible CRT device and reduced ejection fraction

Exclusion Criteria:

* Acute traumatic cardiac injury
* Aortic dissection or aortic root rupture
* Congenital heart diseases such as patent ductus arteriosus, coarctation of aorta, ASD and VSD
* Presence of A-V fistula or intracardiac shunts
* Any contraindications to CMR
* Moderate or severe dysfunction in multiple valves
* Patients with significant claustrophobia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected chronic AS, AR, MR or heart failure with reduced ejection fraction being evaluated for CRT implantation referred for clinically indicated CMR and echocardiography by their cardiologists.. CMR and echocardiography will be clinically indicated in this study group.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-08-23 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in MRI Quantified LVEDVi | 6 months
  10% Change from Baseline - units of measure cc/m2
Change in MRI Quantified LVESVi | 6 months
  15% Change from Baseline - units of measure cc/m2
Change in MRI Quantified LV Strain | 6 months
  5% Change from Baseline
Change in MRI LVEF | 6 Months
  5% Change from Baseline
Change in Kansas City Cardiomyopathy Questionnaire Answers | 6 Months
  Change in quality of life related to heart failure symptoms.
Change in Physical Activity Questionnaire Answers | 6 Months
  Change in physical activity level due to heart failure symptoms.
All-cause mortality | 6 Months
  number of patients expired
Development of class I or IIa indication for valve surgery | 6 Months
  The recommended indications for surgery include: development of symptoms, LV dysfunction (LV end-systolic diameter ≥45 mm or LV ejection fraction ≤60%), and new onset of atrial fibrillation or pulmonary hypertension (systolic pulmonary artery pressure >50 mm Hg at rest).

SECONDARY OUTCOMES:
Accuracy of echocardiography as compared with MRI | 6 Months
  Comparison of MRI measurements based on standard of care echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Kwon, M. D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No